CLINICAL TRIAL: NCT03779087
Title: Efficacies of Two Bismuth Quadruple Therapies in the Second-line Treatment of H Pylori Infection - a Multi-center Randomized Controlled Trial
Brief Title: Efficacies of Two Bismuth Quadruple Therapies in the Second-line Treatment of H Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ping-I (William) Hsu, M.D. (Other)
Responsible Party: Sponsor-Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Organization: Kaohsiung Veterans General Hospital. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS18-CT7-22
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication rate; Rescue treatment
MeSH Terms: interventions — Esomeprazole; Tetracycline; Levofloxacin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10d TL quadruple therapy (Experimental): esomeprazole 40 mg b.i.d. plus tripotassium dicitrate bismuthate 300 mg, tetracycline 500 mg and metronidazole 250 mg q.i.d. for 10 days
  Interventions: Drug: 10d TL quadruple therapy
- 10d AL quadruple therapy (Active Comparator): esomeprazole 40 mg b.i.d. plus tripotassium dicitrate bismuthate 300 mg, amoxicillin 500 mg and metronidazole 250 mg q.i.d. for 10 days
  Interventions: Drug: 10d AL quadruple therapy

INTERVENTIONS:
Drug: 10d TL quadruple therapy — esomeprazole 40 mg bid., tripotassium dicitrate bismuthate 300mg qid, tetracycline 500 mg qid, levofloxacin 500 mg qd.
  Other Names: esomeprazole 40 mg; tripotassium dicitrate bismuthate 300mg; tetracycline 500 mg; levofloxacin 500 mg
  Arms: 10d TL quadruple therapy
Drug: 10d AL quadruple therapy — esomeprazole 40 mg bid., tripotassium dicitrate bismuthate 300mg qid, amoxicillin 500 mg qid, levofloxacin 500 mg qd.
  Other Names: esomeprazole 40 mg; tripotassium dicitrate bismuthate 300mg; amoxicillin 500 mg; levofloxacin 500 mg
  Arms: 10d AL quadruple therapy

SUMMARY:
From the profiles of antibiotic susceptibility data following eradication therapy, tetracycline, amoxicillin and levofloxacin are all good candidates of antibiotics used in the rescue treatment.

DETAILED DESCRIPTION:
The H pylori-infected adult patients with failure of standard triple therapy and H pylori-infected adult patients with failure of non-bismuth quadruple therapy are randomly assigned to either TL quadruple therapy (esomeprazole-bismuth-tetracycline-levofloxacin regimen) or AL quadruple therapy (esomeprazole-bismuth-amoxicillin-levofloxacin regimen) for 10 days. Repeated endoscopy with rapid urease test, histological examination and culture or urea breath tests is performed at six weeks after the end of anti-H pylori therapy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H pylori-infected outpatients, at least 20 years of age with failure of first-line eradication treatments (standard triple, non-bismuth quadruple and bismuth quadruple therapies)

Exclusion Criteria:

* previous allergic reactions to the study medications,
* history of gastrectomy,
* use of antibiotics within the previous 4 weeks,
* pregnant or lactating women,
* coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia, and malignancy).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants in Which H. Pylori Was Eradicated | sixth week after the end of anti- H. pylori therapy
  To assess eradication efficacy,repeated endoscopy with rapid urease test, histological

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan